CLINICAL TRIAL: NCT05312619
Title: The Burden of Lyme Disease (BOLD) in a Pandemic
Brief Title: The Burden of Lyme Disease (BOLD) in a Pandemic - Insights From an Online Cross-sectional and Prospective Cohort Survey
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dr. Daniel Cameron & Associates (Other)
Responsible Party: Principal Investigator, Daniel Cameron, Chief Investigator, Dr. Daniel Cameron & Associates
Other Study IDs: 20212917
Record Dates: First submitted 2022-03-28; First posted 2022-04-05 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: COVID-19; Lyme Disease; COVID-19 Vaccine
MeSH Terms: conditions — COVID-19; Lyme Disease | interventions — Cross-Sectional Studies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Cross sectional survey — A cross-sectional descriptive survey of the Burden of Lyme disease for individual with a history of Lyme disease who contract COVID-19 or are vaccinated against COVID-19

SUMMARY:
A cross-sectional descriptive survey of the BOLD for individuals after having been ill with COVID-19 or have taken the COVID-19 vaccine will be compared with that of individuals who have neither been ill with COVID-19 nor taken the COVID-19 vaccine. Individuals who have both been ill and taken the COVID-19 vaccine will be compared to identify any additive risk factors.

DETAILED DESCRIPTION:
Primary research question:

1. Will the BOLD be worse for individuals who have taken the COVID-19 vaccine?

Secondary research questions:

1. Will the BOLD be worse for individuals who have been ill with COVID-19?
2. What factors affect the BOLD in individuals a) after having been ill with COVID-19, and b) in those who have taken the COVID-19 vaccine? Do they differ?
3. If BOLD risk factors specific to either the COVID-19 vaccine or having been ill with COVID-19 are found, are they additive in people who have experienced both?
4. What is the prevalence of hesitancy in the Lyme disease community to the COVID-19 vaccine?
5. What is the severity of symptoms most likely to predict functional problems in individuals with Lyme disease who have been ill with COVID-19 or taken the COVID-19 vaccine?

ELIGIBILITY:
Inclusion Criteria:

* ≥12 years old
* a self-report of having been diagnosed with Lyme disease.

Exclusion Criteria:

* There are no exclusion criteria.

Min Age: 12 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Individual with a history of Lyme disease who have contracted COVID-19 or have not. Also individual with a history of Lyme disease who have been vaccinated against COVID-19 or have not.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-07-07 (Actual); Primary Completion 2023-07-07 (Estimated); Study Completion 2023-11-07 (Estimated)

PRIMARY OUTCOMES:
Burden of Illness using a General Symptom Questionnaire-30 questionnaire (GSQ-30) | 7/21 to 7/23
  Cross sectional

CONTACTS AND LOCATIONS:
Locations (1):
- Daniel Cameron, Mount Kisco, New York, United States

IPD SHARING:
Plan to Share IPD: No